CLINICAL TRIAL: NCT04785508
Title: Effects Neuromuscular Taping Technique on Upper Limbs Edema in Cardiac Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Antoniucci Maria Enrica, principal investigator, anesthesiology and ICU medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2672
Record Dates: First submitted 2021-02-17; First posted 2021-03-08 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Edema Limbs

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treated group (Experimental): neuromuscolar tape application
  Interventions: Device: neuromuscolar tape
- control group (Active Comparator): antigravity position
  Interventions: Behavioral: antigravity arm position

INTERVENTIONS:
Device: neuromuscolar tape — neuromuscalar tape application in decompression technique (hand and arm)
  Arms: treated group
Behavioral: antigravity arm position — antigravity arm position
  Arms: control group

SUMMARY:
This study aims to verify the efficacy of the decompression technique of neuromuscular taping on cardiac surgery patients in whom edema of the upper limbs occurs due to post-operative water overload.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery patients with postoperative edema of the upper limbs due to water overload

Exclusion Criteria:

* absence of edema,
* previous mastectomy and lymphadenectomy,
* surgery or fractures or infection of the upper limb,
* previous or current deep vein thrombosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
circumference's change of index finger, metacarpus, wrist, mid forearm, elbow and upper arm | measure in millimeter on first postoperative day: before application of tape; and then, every day for the first 3 days, after tape removing, and before the new application.
  measure tissue edema change by circumference change in specific site of the limb ( index finger, metacarpus, wrist, mid forearm, elbow and upper arm)

SECONDARY OUTCOMES:
measurement of the intensity of pain | Measure every day for the 3 days of treatment, before application of tape
  measurement of the intensity of pain during mobilization of fingers, wrist and arm using a VAS scale( 0 is no pain and 10 is the worst possible pain)
movement ability of wrist, hand and arm | measure every day for the 3 days of treatment, before application of tape
  measure angle variation in pronosupination and flexion extension, ulnar and radial deviation of the wrist with articular goniometer
muscle strength measure | measure every day for the 3 days of treatment, before application of tape
  measurement of the handheld gripping force by means of a dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Maria Enrica Antoniucci, MD, Principal Investigator — FPG IRCCS
Locations (1):
- Maria Enrica Antoniucci, Roma, Italy